CLINICAL TRIAL: NCT01621399
Title: A Phase 3, Multicenter, Randomized, Double-blind, Vehicle-controlled Study to Evaluate the Safety and Efficacy of Product 55394 in the Treatment of Bacterial Vaginosis
Brief Title: Safety and Efficacy Study to Treat Bacterial Vaginosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-1601-01
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Treatment with the vehicle (placebo)
  Interventions: Drug: Placebo Vehicle (non-treatment)
- Product 55394 (Experimental): Treatment with product 55394
  Interventions: Drug: Product 55394

INTERVENTIONS:
Drug: Product 55394 — Product 55394 vaginal gel in a prefilled applicator.
  Arms: Product 55394
Drug: Placebo Vehicle (non-treatment) — The vehicle vaginal gel in an applicator (placebo).
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine if product 55394 is safe and efficacious for the treatment of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of bacterial vaginosis as determined by the investigator.
* Other items as identified in the protocol.

Exclusion Criteria:

* Have a known or suspected other infectious cause of vulvovaginitis.
* Other items as identified in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clinical Cure | Day 21
  The proportion of subjects with a clinical cure at the Day 21 visit, as assessed by the investigator.

SECONDARY OUTCOMES:
Therapeutic Cure | Day 21
  The proportion of subjects with a therapeutic cure at the Day 21 visit. Therapeutic cure is defined as both a clinical cure and bacteriological cure as assessed by the investigator and the central laboratory, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Staugaard, Study Director — Medicis Pharmaceutical
Locations (37):
- United States (37):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - La Mesa, California
  - Los Angeles, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Groton, Connecticut
  - Boyton Beach, Florida
  - Clearwater, Florida
  - Miami, Florida
  - North Miami, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Marrero, Louisiana
  - Falls River, Massachusetts
  - Detroit, Michigan
  - Saginaw, Michigan
  - Lincoln, Nebraska
  - Lawrenceville, New Jersey
  - Neptune City, New Jersey
  - Plainsboro, New Jersey
  - Columbus, Ohio
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Jackson, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Schertz, Texas
  - Williston, Vermont
  - Virginia Beach, Virginia
  - Seattle, Washington
  - Tacoma, Washington